CLINICAL TRIAL: NCT03869320
Title: A Single-center, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of ACT-1004-1239 in Healthy Male Subjects (Including Food Interaction, Absolute Bioavailability, Mass Balance, and Metabolite Profiling)
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of ACT-1004-1239 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ID-086-101
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-1004-1239

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, randomized, placebo-controlled, single-ascending dose, Phase 1 study. The food effect will be assessed using a two-period, fixed-sequence design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ACT-1004-1239 (Experimental): ACT-1004-1239 will be given as a single oral dose under fasting conditions. Eight doses are planned with a starting dose of 1 mg. The ADME characteristics and absolute bioavailability using a 14C-radiolabeled microtracer will be evaluated as part of the SAD, after the first 3 cohorts have been performed.
  Interventions: Drug: ACT-1004-1239
- Placebo (Placebo Comparator): Matching placebo will be given as a single oral dose under fasted conditions. Matching placebo for the oral and intravenous administration of the 14C-radiolabeled ACT-1004-1239 will also be available.
  Interventions: Other: Placebo
- Food-effect subpart: ACT-1004-1239 (Experimental): ACT-1004-1239 will be given under both fasted (first period) and fed (second period) conditions. The food effect will be evaluated after the first 3 cohorts have been performed.
  Interventions: Drug: ACT-1004-1239 (Food-effect subpart)
- Food-effect subpart: Placebo (Placebo Comparator): Matching placebo will be given under both fasted (first period) and fed (second period) conditions.
  Interventions: Other: Placebo (Food-effect subpart)

INTERVENTIONS:
Drug: ACT-1004-1239 — ACT-1004-1239 will be available for clinical study use as hard gelatin capsules for oral administration formulated in strengths of 1, 10, and 100 mg. For the ADME subpart, a single oral dose of 1 μCi of 14C radiolabeled ACT-1004-1239 will be given simultaneously with the ACT-1004-1239 capsule. For the absolute bioavailability subpart, a single intravenous dose of a maximum of 1 μCi of 14C radiolabeled ACT-1004-1239 will be given at the expected tmax after the administration of the ACT-1004-1239 capsule.
  Arms: ACT-1004-1239
Other: Placebo — Matching placebo is available as matching capsules for oral administration, formulated with the same excipients but without ACT-1004-1239.
  Arms: Placebo
Drug: ACT-1004-1239 (Food-effect subpart) — ACT-1004-1239 will be available for clinical study use as hard gelatin capsules for oral administration formulated in strengths of 1, 10, and 100 mg.
  Arms: Food-effect subpart: ACT-1004-1239
Other: Placebo (Food-effect subpart) — Matching placebo is available as matching capsules for oral administration, formulated with the same excipients but without ACT-1004-1239.
  Arms: Food-effect subpart: Placebo

SUMMARY:
This Phase 1 study will assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses of ACT-1004-1239 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male subjects aged between 18 and 55 years (inclusive) at Screening.
* No sperm donation from (first) study treatment administration up to at least 90 days after (last) study treatment administration.
* Sexual abstinence or use of condoms from (first) treatment administration up to at least 90 days after (last) study treatment administration. Moreover, the female partner of childbearing potential must use a highly effective method of contraception.

Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Any previous and/or ongoing relevant immune-related disorder or any evidence for immune dysfunction based on medical history and laboratory tests at Screening
* Any cardiac condition or illness (including clinically relevant 12-lead ECG abnormalities) with a potential to increase the cardiac risk of the subject based on medical history and 12-lead ECG measured at Screening.
* QT interval corrected with Fridericia's formula (QTcF) > 430 ms, respectively, QRS interval > 110 ms, PR interval > 200 ms, or heart rate (HR) > 90 bpm on 12-lead ECG at Screening and Day 1 pre-dose (of the first period when applicable).
* Treatment with another investigational treatment within the 2 months prior to Screening or participation in more than 3 investigational treatment studies within the year prior to Screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition that might interfere with the ADME of the study treatment (e.g., appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Previous treatment with any prescribed medications (including vaccines and strong CYP3A4 inhibitors/inducers) or over-the-counter (OTC) medications (including homeopathic preparations, herbal medicines, vitamins, and minerals) within the 2 weeks or 5 terminal half-lives (t½; whichever is longer) prior to (first) study treatment administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent (serious) adverse events (AEs and SAEs) | From baseline up to EOS of each cohort (total duration: up to 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Pharmaron CPC, Inc. & Affiliates, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huynh C, Seeland S, Segrestaa J, Gnerre C, Hogeback J, Meyer Zu Schwabedissen HE, Dingemanse J, Sidharta PN. Absorption, Metabolism, and Excretion of ACT-1004-1239, a First-In-Class CXCR7 Antagonist: In Vitro, Preclinical, and Clinical Data. Front Pharmacol. 2022 Mar 30;13:812065. doi: 10.3389/fphar.2022.812065. eCollection 2022. PMID 35431953
- [Derived] Pouzol L, Baumlin N, Sassi A, Tunis M, Marrie J, Vezzali E, Farine H, Mentzel U, Martinic MM. ACT-1004-1239, a first-in-class CXCR7 antagonist with both immunomodulatory and promyelinating effects for the treatment of inflammatory demyelinating diseases. FASEB J. 2021 Mar;35(3):e21431. doi: 10.1096/fj.202002465R. PMID 33595155